CLINICAL TRIAL: NCT01900405
Title: Intranasal Dexmedetomidine Sedation for Pediatric Computerized Tomography Imaging
Brief Title: Intranasal Dexmedetomidine Sedation for Pediatric CT Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Eduardo Mekitarian Filho, MD, MsC, PhD, University of Sao Paulo
Other Study IDs: USPDex
Record Dates: First submitted 2013-07-09; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Traumatic Brain Injury; Children
Keywords: Dexmedetomidine; Administration, Intranasal; Children; Computerized Tomography
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dexmedetomidine: All children undergoing
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex (brand name)

SUMMARY:
This study has the objective to determine if intranasal dexmedetomidine, a sedative, is suitable for pediatric sedation in children undergoing tomographic scans.

DETAILED DESCRIPTION:
Invasive procedures for diagnosis in children are a routine part of an emergency care department. Most of these procedures are painful and uncomfortable for both the child and for their families, and impossible to be performed without patient immobilization. Thus, procedural sedation is critical to this end. Procedural sedation can be defined as the use of sedatives, analgesics, or dissociative drugs for anxiolysis, analgesia, sedation and motor control during painful procedures.

The increasing demand of pediatric emergency services and, consequently, the performance of procedures that require sedation, made it impossible for universal coverage of anesthesiologists in such procedures. As a result, a wide variety of drugs, sedation techniques and different degrees of effectiveness and adverse effects of sedation, such as irritability and sedation failure are described.

Particularly in children who need CT scan, there is usually no need for venous access for sedation. However, our most used drug, chloral hydrate, was abandoned in most centers outside the country. When administered orally, the drug produces malaise and vomiting, and gastric mucosal irritation, in addition, the rectal absorption is unpredictable. Additionally, in recent years increasing importance has been given to the fact that the drug be related, in vitro, the increased carcinogenicity in mice by cellular structural change, which is leading to the ban of same drug in the United States and in some european countries.

Dexmedetomidine is a highly selective alpha-2 agonist receptors, which has the advantage of mimicking natural sleep, according to electroencephalographic studies, with low incidence of adverse events. Its application as a sedative in pediatric procedures, as well as pre-anesthetic medication, has been increasingly described according to recent studies. The intranasal route has been used with the advantage of avoiding a venous line or intramuscular injection, with good results; however, it hasn't been described yet in children undergoing CT scans.

Thus, this work is justified to describe, in a pioneering way, the use of intranasal dexmedetomidine for sedation for CT, documenting its efficacy and safety in a specific cohort of patients sedated for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 month to 15 years old undergoing CT scans in the pediatric emergency department

Exclusion Criteria:

* Glasgow coma scale < 13
* Epistaxis or suspected base skull fracture
* Use of contrast or need for an IV line before sedation
* Uncontrolled gastroesophageal reflux or vomiting
* Current (or within past 3 months) history of apnea of prematurity requiring an apnea monitor
* Acute, unstable respiratory disease
* Unstable cardiac status
* Craniofacial anomaly
* Medication use: digoxin
* Moya Moya Disease
* New onset stroke
* American Society of Anesthesiologists physical status ≥3

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The University Hospital of University of Sao Paulo is a secondary teaching hospital. The Pediatric Emergency Department has over 6,000 consultations per month, mainly in children without underlying diseases. Respiratory diseases are the leading causes of hospital admission. During the study period, any children presented to the emergency department with indication for a CT scanning will be recruited for IN dexmedetomidine, respecting the exclusion criteria displayed below.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Rates of sedation failure with intranasal dexmedetomidine for sedation for pediatric CT imaging | Failure to sedate will be defined as non-completion of CT imaging after 2 nasal doses of dexmedetomidine (2.5 mcg/kg at admission; 0.5 mcg/kg after 15 minutes if not sedated).
  Main outcome for this research is to know if IN dexmedetomidine is effective for adequate sedation in children undergoing CT scannings. This will be reported as percentage of failed sedations, if they occur. Failed sedations will be defined if after a initial 2.5 mcg/kg dose along with another 0.5 mcg/kg dose after 15 minutes, the child does not sedate.

SECONDARY OUTCOMES:
Safety of IN dexmedetomidine for pediatric CT imaging | At admission and every 5 minutes after sedation
  Patients will be fully monitored every five minutes after IN dexmedetomidine administration, with heart rate, respiratory rate, non-invasive blood pressure and pulse oximetry. Any adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Keira Mason, MD, Study Director — Boston Children's Hospital, Harvard Medical School
Locations (1):
- University Hospital, University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mekitarian Filho E, Robinson F, de Carvalho WB, Gilio AE, Mason KP. Intranasal dexmedetomidine for sedation for pediatric computed tomography imaging. J Pediatr. 2015 May;166(5):1313-1315.e1. doi: 10.1016/j.jpeds.2015.01.036. Epub 2015 Mar 6. PMID 25748567